CLINICAL TRIAL: NCT06458426
Title: Thermoregulation in Individuals With a Leg Amputation: Mechanics and Vascular Physiology Factors to Understand Risks for Tissue Complications
Brief Title: Thermoregulation in Individuals With a Leg Amputation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Kota Takahashi, Assistant Professor, University of Utah
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00155345
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Amputation; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rigid Pylon (Experimental): The prosthesis will be given a commercial prosthetic foot and a rigid pylon that connects the prosthetic foot to the socket.
  Interventions: Device: shock-absorbing prosthesis
- Shock-absorbing Pylon (Experimental): The prosthesis will be given a commercial prosthetic foot and a compressive 'shock-absorbing' pylon that connects the prosthetic foot to the socket.
  Interventions: Device: shock-absorbing prosthesis

INTERVENTIONS:
Device: shock-absorbing prosthesis — the intervention will test the difference between rigid and shock-absorbing pylons, while the same prosthetic foot is applied in each condition.

SUMMARY:
The goal of this project is to understand the factors that affect skin temperature (e.g., tissue above amputation site, and opposite foot) in people with amputation and diabetes. This project will also test the effects of 'shock-absorbing' prosthesis on skin temperature responses.

DETAILED DESCRIPTION:
The overall goal of this project is to understand the factors that affect impaired temperature control in individuals with a leg amputation for areas vulnerable to damage, such as the tissue above the amputation site and the opposite intact foot. Abnormal tissue temperature is associated with risks for tissue damage, such as ulcers and pressure sores, especially in people with diabetes. In this study, we aim to study the effects of biomechanics and vascular physiology on tissue temperature responses. We will also determine the effectiveness of prosthetic shock-absorbing components in protecting the tissue from damage.

It is hypothesized that the temperatures of tissues above the amputation site and in the opposite intact foot are associated with mechanical factors during walking, such as shear forces and work (i.e., energy). It is also hypothesized that impaired temperature regulation, especially in people with diabetes, is associated with poor vascular function that inhibits effective blood circulation and oxygen delivery to affected tissues. Lastly, it is hypothesized that walking with a shock-absorbing prosthetic component can improve comfort and improve temperature regulation of tissues above the amputation site.

This project will recruit 40 individuals with a unilateral transtibial (below-knee) amputation, divided into two groups: with and without diabetes. All individuals will be given two sets of prostheses: with and without a shock-absorbing pylon (SAP). SAP is a modular prosthetic component that connects the socket and the foot components and allows added compression and twisting along the pylon. In both sets of prostheses conditions, the participants will wear the same foot component provided by the research team. For each of the two sets of prostheses (with and without SAP), the participants will make up to 5 visits to the laboratory (i.e., up to 10 total visits for the entire protocol). Each visit will involve data collections under a variety of walking tasks, such as walking on various slopes and turning. The same data collections will be repeated with the other set of prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a unilateral transtibial amputation, divided into two groups (with and without diabetes)
* Participants must classify as Medicare class K2 or higher (who can traverse low-level environmental barriers such as curbs, stairs or uneven surfaces).
* Participants must have undergone amputation at least 6 months prior.
* They must have the ability to walk for at least 10 continuous minutes without undue fatigue.

Exclusion Criteria:

* Neurological impairment that may affect walking function, such as stroke, severe traumatic brain injury, Parkinson's disease, and multiple sclerosis.
* History of inflammatory diseases, such as Raynaud's syndrome or rheumatoid arthritis.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Walking mechanics | during the intervention/procedure/surgery
  Mechanics of walking will be collected using a high-speed motion capture system and force-sensing platforms, which will quantify the motion of the legs and forces acting on the legs, respectively.
Vascular physiology - macrocirculation | during the intervention/procedure/surgery
  Macrocirculation of the legs (i.e.,blood flow) will be recorded using a Doppler ultrasound probe secured over the thigh during walking
Vascular physiology - microcirculation | during the intervention/procedure/surgery
  Microcirculation of the legs (i.e.,oxygen utility) will be recorded using near-infrared spectroscopy sensors placed on the thighs, calf, and top surface of the foot.
Temperature in lower limb | during the intervention/procedure/surgery
  Temperatures of the skin above the amputation site and the opposite intact foot will be recorded using thermistors and a thermal imaging camera.
Comfort | during the intervention/procedure/surgery
  Participants will complete a self-reported questionnaire to indicate comfort while walking with a prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Kota Takahashi, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No